CLINICAL TRIAL: NCT00003048
Title: Phase II Study of Intravenous Amifostine in Myelodysplastic Syndrome
Brief Title: Amifostine in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DM97-041; P30CA016672 (NIH); MDA-DM-97-041 (Other: UT MD Anderson Cancer Center); ALZA-97-007-ii; ALZA-MDA-DM-97-041; NCI-V97-1300; CDR0000065687 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-09-06 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; Amifostine; Ethyol; Ethiofos; Gammaphos
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Amifostine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amifostine (Experimental): Amifostine IV 2 weeks, followed by 2 weeks rest (4 week cycle)
  Interventions: Drug: Amifostine Trihydrate

INTERVENTIONS:
Drug: Amifostine Trihydrate — Escalating dose IV for two weeks, followed by 2 weeks of rest. Each treatment cycle is 4 weeks.
  Other Names: Ethyol; Ethiofos; Gammaphos

SUMMARY:
RATIONALE: Amifostine may improve blood counts in patients with myelodysplastic syndrome.

PURPOSE: Phase II trial to study the effectiveness of amifostine in treating patients with myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Define the activity of amifostine in improving blood counts in patients with myelodysplastic syndrome.

OUTLINE: This is an open label, nonrandomized, single center, dose escalation study. Patients receive amifostine IV for two weeks, followed by 2 weeks of rest. Each treatment cycle is 4 weeks. Responses are evaluated after each cycle (for a minimum of 2 induction cycles). Patients with a grade 0 toxicity in the first course receive a 25% increase in dose during the second course. Patients with grade 1 or 2 toxicity receive no dose change. Patients with grade 3 toxicity receive a 25% reduction in dose or treatment is stopped. All patients demonstrating response are eligible for maintenance therapy. Treatment is continued for up to 12 months or a total of 13 cycles.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven myelodysplastic syndrome Less than 30% blasts in bone marrow

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: Zubrod 0-2 Karnofsky 60-100% ECOG 0-2 Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2 mg/dL Renal: Creatinine no greater than 2 mg/dL Cardiovascular: No New York Heart Association Class IV disease No antihypertensive medication within 24 hours of amifostine administration Other: Not pregnant or nursing Effective contraceptive method must be used during study No medical illness No psychosis Eligible patients with an HLA compatible donor are referred to bone marrow transplantation

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy within 4 weeks of study and recovered Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 1997-06-05; Primary Completion 2001-02-12 (Actual); Study Completion 2001-02-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Amifostine | After each 4 week cycle
  Responses are evaluated after each cycle (for a minimum of 2 induction cycles).

CONTACTS AND LOCATIONS:
Overall Officials: Razelle Kurzrock, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org